CLINICAL TRIAL: NCT00005301
Title: Transfusion Safety Study (TSS)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 3002
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2001-08

CONDITIONS: Acquired Immunodeficiency Syndrome; Blood Transfusion; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

SUMMARY:
To evaluate factors influencing the risk of transfusion-transmitted human immunodeficiency virus (HIV) infection and its progression to clinically significant manifestations.

DETAILED DESCRIPTION:
BACKGROUND:

In the summer of 1981, the Centers for Disease Control (CDC) alerted the medical community to an unexpected outbreak of Pneumocystis carinii pneumonia and Kaposi's sarcoma in young homosexual men, individuals not known to be at risk for these uncommon diseases. Studies of immunologic functions in these patients demonstrated lymphopenia, cutaneous anergy, reduced helper T-lymphocyte (T4) subpopulations, depressed ratios of helper T-lymphocytes to suppressor T-lymphocytes (T4:T8), abnormal lymphocyte responses to mitogen stimulation, decreased natural killer-cell activity, and often hypergammaglobulinemia. The name of acquired immunodeficiency syndrome (AIDS) was given to this disorder of immunologic regulation with opportunistic infections or Kaposi's sarcoma or both.

Since that time, AIDS was reported in patients with hemophilia and in others receiving blood transfusions. The NHLBI was delegated responsibility for studies to elucidate, through a systematic prospective study, the possible association of blood product use with AIDS. The incidence of transfusion-acquired AIDS was so low as to preclude a general prospective study of transfusion recipients to determine the overall incidence of the disease. By focusing on patient groups that appeared to have a higher likelihood for developing AIDS because they required chronic, repeated transfusion therapy, information about the epidemiology of the disorder could be more readily obtained. Continuing medical evaluation of these patients from apparent high-risk groups in a prospective fashion allowed identification of significant emerging physiologic alterations and to follow the time-course of pathologic developments.

The purpose of this study was to develop a clear picture of what immunologic changes occurred in patients who were transfused and to determine when these changes occurred and how long they lasted. Since most of the patient population was heavily transfused, some of the study subjects eventually developed AIDS. Information obtained during the study about these patients was then used to answer such questions as: Which factors determined a particular person's risk of developing AIDS and to what degree? What alterations occurred before the clinical manifestations of AIDS? Was progression from normal to defective cell-mediated immunity to AIDS strictly unidirectional or did altered cell-mediated immunity in the study cohort ever regress to normality? If progression was not unidirectional, what determined the outcome? Also, the importance of establishing a serum and cell repository could not be overemphasized, since, as new scientific information became available, these specimens enabled the performance of a number of different retrospective studies.

In 1984 a serum repository for HIV testing was established. The task of the repository was to collect and store serum samples from blood donors in four blood transfusion units located in four major risk areas for AIDS, namely New York, San Francisco, Miami, and Los Angeles. Blood was obtained from the New York Blood Center in New York City, the Irwin Memorial Blood Bank in San Francisco, the Red Cross in Los Angeles, and the American Red Cross, South Florida Region, in Miami. The purpose of the repository was to determine the outcome of the transfusion of blood components retrospectively found to show HIV infection of the donor. The collected sera were separated, indexed, frozen, and stored.

In 1984 the second part of the Transfusion Safety Study, the prospective study, was initiated by NHLBI under a separate request for proposal. The testing of the 201,000 serum specimens in the donor repository for antibody to HIV was carried out by laboratories in the prospective study. Those donors confirmed to be anti-HIV positive and matching donors confirmed to be anti-HIV negative were recruited as TSS subjects. Recipients of blood from the positive donors and the negative donors were also recruited as subjects.

In September 1984, the TSS began a nine month planning phase during which the protocols and data systems for the prospective study were developed. Subjects were entered in July 1985 through June 1989. Analysis continued through November 1997. There were clinical centers in Los Angeles, San Francisco, New York City, and Miami. The coordinating center was at the University of Southern California. The central laboratories including the immunological standardization laboratory, the immunological reagents laboratory, and the central processing laboratory were located in Los Angeles, with one of the immunology laboratories located in Seattle, Washington at the Puget Sound Blood Center.

DESIGN NARRATIVE:

At baseline, each subject received a physical examination, was questioned as to medical history, and gave blood samples for immunologic and other studies. Each subject returned at a specified interval for a repeat of studies specified in the protocol. Blood studies included complete blood cell count, characterization of immunologic cells such as T- and B-lymphocytes and natural killer-cells. Plasma and Buffy coat cell suspensions were stored frozen. Alanine aminotransferase levels were determined. Serologic tests were performed for hepatitis, Epstein-Barr virus, and cytomegalovirus. Markers of immune status, including immune globulin levels were measured. The study ended in November, 1997.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1984-09; Study Completion 1998-02

CONTACTS AND LOCATIONS:
Overall Officials: James Mosley

REFERENCES:
- [Background] Niland-Weiss J, Azen SP, Odom-Maryon T, Lui F, Hagerty C. A microcomputer-based distributed data management system for a large cooperative study of transfusion associated acquired immunodeficiency syndrome. Comput Biomed Res. 1987 Jun;20(3):225-43. doi: 10.1016/0010-4809(87)90056-5. PMID 3608439
- [Background] Fletcher MA, Baron GC, Ashman MR, Fischl MA, Klimas NG. Use of whole blood methods in assessment of immune parameters in immunodeficiency states. Diagn Clin Immunol. 1987;5(2):69-81. PMID 3113759
- [Background] Perkins HA, Cordell R, Bueno C, Shiota J, Hitchcock B. The progressive decrease in the proportion of blood donors with antibody to the human immunodeficiency virus (HIV). Transfusion. 1987 Nov-Dec;27(6):502-3. doi: 10.1046/j.1537-2995.1987.27688071706.x. No abstract available. PMID 3686662
- [Background] Kaplan J, Sarnaik I, Lusher J. Increase in Leu 2+ Leu 7+ lymphocytes in HIV 1-seropositive patients with hemophilia repeatedly treated with clotting factor concentrates. Clin Immunol Immunopathol. 1988 Mar;46(3):337-41. doi: 10.1016/0090-1229(88)90052-9. PMID 3257429
- [Background] Brown NA, Kovacs A, Lui CR, Hur C, Zaia JA, Mosley JW. Prevalence of antibody to human herpesvirus 6 among blood donors infected with HIV. Lancet. 1988 Nov 12;2(8620):1146. doi: 10.1016/s0140-6736(88)90570-3. No abstract available. PMID 2903363
- [Background] Aledort LM. Blood products and immune changes: impacts without HIV infection. Semin Hematol. 1988 Apr;25(2 Suppl 1):14-9. No abstract available. PMID 3133772
- [Background] Bishop PC, Boone D, Parker JW. Immunophenotypes by flow cytometry: a longitudinal study in healthy individuals. Diagn Clin Immunol. 1988;5(5):232-40. PMID 3359565
- [Background] Gjerset GF, Vyas GN, Bhat R, Operskalski EA. Phenotypes for group-specific component among patients exposed to human immunodeficiency virus by transfusions. J Infect Dis. 1988 Mar;157(3):609-10. doi: 10.1093/infdis/157.3.609. No abstract available. PMID 3343536
- [Background] Govindarajan S, Edwards VM, Stuart ML, Operskalski EA, Mosley JW and the Transfusion Safety Study Group: Influence of Human Immunodeficiency Virus Infection Upon Expression of Chronic Hepatitis B and D Virus Infections. In: Zuckerman AJ (Ed), Viral Hepatitis and Liver Disease, Alan R Liss, Inc, New York, pp 210-214, 1988
- [Background] McClure E, Gaynor S, Veiga-Benach A, O'Neil D, and the Transfusion Safety Study Group: Notification of Recipients of Human Immunodeficiency Virus (HIV) Antibody Positive Transfusions. Nursing, Jan; 10, 1989
- [Background] Norman GL, Barker SS, Rasheed S. Immunoblot reactivity of a non-HIV protein with human sera. Transfusion Safety Study Group. J Clin Lab Anal. 1989;3(3):148-51. doi: 10.1002/jcla.1860030303. PMID 2787852
- [Background] Mosley JW, Nowicki M, Kleinman SH, Dietrich SL and the Transfusion Safety Study Group: Reactivation of Hepatitis B. Lancet, 1:1083-1084, 1989
- [Background] Fletcher MA, Azen SP, Adelsberg B, Gjerset G, Hassett J, Kaplan J, Niland JC, Odom-Maryon T, Parker JW, Stites DP, et al. Immunophenotyping in a multicenter study: the Transfusion Safety Study experience. Clin Immunol Immunopathol. 1989 Jul;52(1):38-47. doi: 10.1016/0090-1229(89)90191-8. PMID 2656018
- [Background] Kleinman SH, Niland JC, Azen SP, Operskalski EA, Barbosa LH, Chernoff AI, Edwards VM, Lenes BA, Marshall GJ, Nemo GJ, et al. Prevalence of antibodies to human immunodeficiency virus type 1 among blood donors prior to screening. The Transfusion Safety Study/NHLBI Donor Repository. Transfusion. 1989 Sep;29(7):572-80. doi: 10.1046/j.1537-2995.1989.29789369672.x. PMID 2672433
- [Background] Lang DJ, Kovacs AA, Zaia JA, Doelkin G, Niland JC, Aledort L, Azen SP, Fletcher MA, Gauderman J, Gjerset GJ, et al. Seroepidemiologic studies of cytomegalovirus and Epstein-Barr virus infections in relation to human immunodeficiency virus type 1 infection in selected recipient populations. Transfusion Safety Study Group. J Acquir Immune Defic Syndr (1988). 1989;2(6):540-9. PMID 2555471
- [Background] Operskalski EA, Schiff ER, Kleinman SH, Busch M, Taylor PE, Parks WP, Lee H, Tomasulo PA, Donegan E, Stuart M, et al. Epidemiologic background of blood donors with antibody to human T-cell lymphotropic virus. Transfusion Safety Study Group. Transfusion. 1989 Oct;29(8):746-8. doi: 10.1046/j.1537-2995.1989.29890020448.x. PMID 2572078
- [Background] Edwards VM, Mosley JW. Reproducibility in quality control of protein (Western) immunoblot assay for antibodies to human immunodeficiency virus. Am J Clin Pathol. 1989 Jan;91(1):75-8. doi: 10.1093/ajcp/91.1.75. PMID 2910017
- [Background] Parker JW, Adelsberg B, Azen SP, Boone D, Fletcher MA, Gjerset GF, Hassett J, Kaplan J, Niland JC, Odom-Maryon T, et al. Leukocyte immunophenotyping by flow cytometry in a multisite study: standardization, quality control, and normal values in the Transfusion Safety Study. The Transfusion Safety Study Group. Clin Immunol Immunopathol. 1990 May;55(2):187-220. doi: 10.1016/0090-1229(90)90097-a. PMID 2182228
- [Background] Donegan E, Busch MP, Galleshaw JA, Shaw GM, Mosley JW. Transfusion of blood components from a donor with human T-lymphotropic virus type II (HTLV-II) infection. The Transfusion Safety Study Group. Ann Intern Med. 1990 Oct 1;113(7):555-6. doi: 10.7326/0003-4819-113-7-555. No abstract available. PMID 2393211
- [Background] Busch MP, Donegan E, Stuart M, Mosley JW. Donor HIV-1 p24 antigenaemia and course of infection in recipients Transfusion Safety Study Group. Lancet. 1990 Jun 2;335(8701):1342. doi: 10.1016/0140-6736(90)91221-u. No abstract available. PMID 1971398
- [Background] Busch MP, Taylor PE, Lenes BA, Kleinman SH, Stuart M, Stevens CE, Tomasulo PA, Allain JP, Hollingsworth CG, Mosley JW. Screening of selected male blood donors for p24 antigen of human immunodeficiency virus type 1. The Transfusion Safety Study Group. N Engl J Med. 1990 Nov 8;323(19):1308-12. doi: 10.1056/NEJM199011083231904. PMID 2120588
- [Background] Dietrich SL, Mosley JW, Lusher JM, Hilgartner MW, Operskalski EA, Habel L, Aledort LM, Gjerset GF, Koerper MA, Lewis BH, et al. Transmission of human immunodeficiency virus type 1 by dry-heated clotting factor concentrates. Transfusion Safety Study Group. Vox Sang. 1990;59(3):129-35. doi: 10.1111/j.1423-0410.1990.tb00846.x. PMID 2124751
- [Background] Donegan E, Stuart M, Niland JC, Sacks HS, Azen SP, Dietrich SL, Faucett C, Fletcher MA, Kleinman SH, Operskalski EA, et al. Infection with human immunodeficiency virus type 1 (HIV-1) among recipients of antibody-positive blood donations. Ann Intern Med. 1990 Nov 15;113(10):733-9. doi: 10.7326/0003-4819-113-10-733. PMID 2240875
- [Background] Busch MP, Young MJ, Samson SM, Mosley JW, Ward JW, Perkins HA. Risk of human immunodeficiency virus (HIV) transmission by blood transfusions before the implementation of HIV-1 antibody screening. The Transfusion Safety Study Group. Transfusion. 1991 Jan;31(1):4-11. doi: 10.1046/j.1537-2995.1991.31191096183.x. PMID 1986462
- [Background] Parks WP, Lenes BA, Tomasulo PA, Schiff ER, Parks ES, Shaw GM, Lee H, Yan HQ, Lai S, Hollingsworth CG, et al. Human T-cell lymphotropic virus infection among blood donors in south Florida. The Transfusion Safety Study Group. J Acquir Immune Defic Syndr (1988). 1991;4(1):89-96. PMID 1670589
- [Background] Aledort LM, Hilgartner MW, Pike MC, Gjerset GF, Koerper MA, Lian EY, Lusher JM, Mosley JW. Variability in serial CD4 counts and relation to progression of HIV-I infection to AIDS in haemophilic patients. Transfusion Safety Study Group. BMJ. 1992 Jan 25;304(6821):212-6. doi: 10.1136/bmj.304.6821.212. PMID 1346752
- [Background] Busch MP, Henrard DR, Hewlett IK, Mehaffey WF, Epstein JS, Allain JP, Lee TH, Mosley JW. Poor sensitivity, specificity, and reproducibility of detection of HIV-1 DNA in serum by polymerase chain reaction. The Transfusion Safety Study Group. J Acquir Immune Defic Syndr (1988). 1992;5(9):872-7. PMID 1512686
- [Background] Fletcher MA, Mosley JW, Hassett J, Gjerset GF, Kaplan J, Parker JW, Donegan E, Lusher JM, Lee H. Effect of age on human immunodeficiency virus type 1-induced changes in lymphocyte populations among persons with congenital clotting disorders. Transfusion Safety Study Group. Blood. 1992 Aug 1;80(3):831-40. PMID 1638032
- [Background] Donegan E, Pell P, Lee H, Shaw GM, Mosley JW. Transmission of human T-lymphotropic virus type I by blood components from a donor lacking anti-p24: a case report. The Transfusion Safety Study Group. Transfusion. 1992 Jan;32(1):68-71. doi: 10.1046/j.1537-2995.1992.32192116436.x. PMID 1731439
- [Background] Fletcher MA, Gjerset GF, Hassett J, Donegan E, Parker JW, Mosley JW. Lymphocyte immunophenotypes among anti-HTLV-I/II-positive blood donors and recipients. The Transfusion Safety Study Group. J Acquir Immune Defic Syndr (1988). 1991;4(6):628-32. PMID 1673714
- [Background] Buckley JD, Pike MC, Mosley JW. Statistical approaches to evaluating prognostic indices in HIV infection. The Transfusion Safety Study Group. AIDS. 1991 Nov;5(11):1398. doi: 10.1097/00002030-199111000-00027. No abstract available. PMID 1768396
- [Background] Odom-Maryon T, Langholz B, Niland J, Azen S. Generalization of normal discriminant analysis using Fourier series density estimators. Transfusion Safety Study Group. Stat Med. 1991 Mar;10(3):473-85. doi: 10.1002/sim.4780100319. PMID 2028130
- [Background] Miller K, Donegan E, Curran P, Shelley TJ. Effects of counselling on knowledge about HIV-1 among transfusion recipients and their partners. Transfusion Safety Study Group. AIDS Care. 1990;2(2):155-62. doi: 10.1080/09540129008257726. PMID 2085537
- [Background] Operskalski EA, Stram DO, Lee H, Zhou Y, Donegan E, Busch MP, Stevens CE, Schiff ER, Dietrich SL, Mosley JW. Human immunodeficiency virus type 1 infection: relationship of risk group and age to rate of progression to AIDS. Transfusion Safety Study Group. J Infect Dis. 1995 Sep;172(3):648-55. doi: 10.1093/infdis/172.3.648. PMID 7658055
- [Background] Diaz RS, Sabino EC, Mayer A, Mosley JW, Busch MP. Dual human immunodeficiency virus type 1 infection and recombination in a dually exposed transfusion recipient. The Transfusion Safety Study Group. J Virol. 1995 Jun;69(6):3273-81. doi: 10.1128/JVI.69.6.3273-3281.1995. PMID 7745674
- [Background] Wong WY, Powars DR, Operskalski EA, Hassett J, Parker JW, Sarnaik S, Pegelow CH, Hilgartner MW, Johnson CS, Zhou Y, et al. Blood transfusions and immunophenotypic alterations of lymphocyte subsets in sickle cell anemia. The Transfusion Safety Study Group. Blood. 1995 Apr 15;85(8):2091-7. PMID 7718880
- [Background] Busch MP, Operskalski EA, Mosley JW, Stevens CE, Schiff ER, Kleinman SH, Lee H, Lee M, Harris M. Epidemiologic background and long-term course of disease in human immunodeficiency virus type 1-infected blood donors identified before routine laboratory screening. Transfusion Safety Study Group. Transfusion. 1994 Oct;34(10):858-64. doi: 10.1046/j.1537-2995.1994.341095026970.x. PMID 7940656
- [Background] Hilgartner M. Results of the transfusion safety study. Ann Hematol. 1994;68 Suppl 3:S59. doi: 10.1007/BF01774536. No abstract available. PMID 7910043
- [Background] Hilgartner MW. Changes in CD4 count relative to product usage: findings from the transfusion safety study. Semin Hematol. 1993 Oct;30(4 Suppl 5):7-9. No abstract available. PMID 7903481
- [Background] Hilgartner MW, Buckley JD, Operskalski EA, Pike MC, Mosley JW. Purity of factor VIII concentrates and serial CD4 counts. The Transfusion Safety Study Group. Lancet. 1993 May 29;341(8857):1373-4. doi: 10.1016/0140-6736(93)90943-b. PMID 8098792
- [Background] Mosley JW. Low CD4+ counts in a study of transfusion safety: correction. N Engl J Med. 1993 Apr 15;328(15):1128. doi: 10.1056/NEJM199304153281515. No abstract available. PMID 8096065
- [Background] Aledort LM, Operskalski EA, Dietrich SL, Koerper MA, Gjerset GF, Lusher JM, Lian EC, Mosley JW. Low CD4+ counts in a study of transfusion safety. The Transfusion Safety Study Group. N Engl J Med. 1993 Feb 11;328(6):441-2. doi: 10.1056/NEJM199302113280614. No abstract available. PMID 8093638
- [Background] Mosley JW, Nowicki MJ, Kasper CK, Donegan E, Aledort LM, Hilgartner MW, Operskalski EA. Hepatitis A virus transmission by blood products in the United States. Transfusion Safety Study Group. Vox Sang. 1994;67 Suppl 1:24-8. PMID 8091731
- [Background] Hassett J, Gjerset GF, Mosley JW, Fletcher MA, Donegan E, Parker JW, Counts RB, Aledort LM, Lee H, Pike MC. Effect on lymphocyte subsets of clotting factor therapy in human immunodeficiency virus-1-negative congenital clotting disorders. The Transfusion Safety Study Group. Blood. 1993 Aug 15;82(4):1351-7. PMID 8353293
- [Background] Adams M, Lee TH, Busch MP, Heitman J, Marshall GJ, Gjerset GF, Mosley JW. Rapid freezing of whole blood or buffy coat samples for polymerase chain reaction and cell culture analysis: application to detection of human immunodeficiency virus in blood donor and recipient repositories. The Transfusion Safety Study Group. Transfusion. 1993 Jun;33(6):504-8. doi: 10.1046/j.1537-2995.1993.33693296814.x. PMID 8516793
- [Background] Operskalski EA, Busch MP, Mosley JW, Stram DO. Comparative rates of disease progression among persons infected with the same or different HIV-1 strains. The Transfusion Safety Study Group. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Jun 1;15(2):145-50. doi: 10.1097/00042560-199706010-00008. PMID 9241114
- [Background] Operskalski EA, Mosley JW, Busch MP, Stram DO. Influences of age, viral load, and CD4+ count on the rate of progression of HIV-1 infection to AIDS. Transfusion Safety Study Group. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Jul 1;15(3):243-4. doi: 10.1097/00042560-199707010-00009. No abstract available. PMID 9257660
- [Background] Wong WY, Zhou Y, Operskalski EA, Hassett J, Powars DR, Mosley JW. Hematologic profile and lymphocyte subpopulations in hemoglobin SC disease: comparison with hemoglobin SS and black controls. The Transfusion Safety Study Group. Am J Hematol. 1996 Jul;52(3):150-4. doi: 10.1002/1096-8652(199607)52:33.0.co;2-6. PMID 8756079
- [Background] Busch MP, Operskalski EA, Mosley JW, Lee TH, Henrard D, Herman S, Sachs DH, Harris M, Huang W, Stram DO. Factors influencing human immunodeficiency virus type 1 transmission by blood transfusion. Transfusion Safety Study Group. J Infect Dis. 1996 Jul;174(1):26-33. doi: 10.1093/infdis/174.1.26. PMID 8656010
- [Background] Kedes DH, Operskalski E, Busch M, Kohn R, Flood J, Ganem D. The seroepidemiology of human herpesvirus 8 (Kaposi's sarcoma-associated herpesvirus): distribution of infection in KS risk groups and evidence for sexual transmission. Nat Med. 1996 Aug;2(8):918-24. doi: 10.1038/nm0896-918. PMID 8705863
- [Background] Gjerset GF, Pike MC, Mosley JW, Hassett J, Fletcher MA, Donegan E, Parker JW, Counts RB, Zhou Y, Kasper CK, et al. Effect of low- and intermediate-purity clotting factor therapy on progression of human immunodeficiency virus infection in congenital clotting disorders. Transfusion Safety Study Group. Blood. 1994 Sep 1;84(5):1666-71. PMID 7915149
- [Background] Diaz RS, Zhang L, Busch MP, Mosley JW, Mayer A. Divergence of HIV-1 quasispecies in an epidemiologic cluster. AIDS. 1997 Mar 15;11(4):415-22. doi: 10.1097/00002030-199704000-00003. PMID 9084787
- [Background] Zhang L, Diaz RS, Ho DD, Mosley JW, Busch MP, Mayer A. Host-specific driving force in human immunodeficiency virus type 1 evolution in vivo. J Virol. 1997 Mar;71(3):2555-61. doi: 10.1128/JVI.71.3.2555-2561.1997. PMID 9032400
- [Background] Diaz RS, Sabino EC, Mayer A, deOliveira CF, Mosley JW, Busch MP. Lack of dual HIV infection in a transfusion recipient exposed to two seropositive blood components. AIDS Res Hum Retroviruses. 1996 Sep 1;12(13):1291-5. doi: 10.1089/aid.1996.12.1291. No abstract available. PMID 8870851
- [Background] Mosley JW. Has hepatitis A virus been transmitted by clotting factor concentrates among hemophiliacs in the United States? Vox Sang. 1994;67 Suppl 4:12-5; discussion 24-6. PMID 7831863
- [Background] Operskalski EA, Stram DO, Busch MP, Huang W, Harris M, Dietrich SL, Schiff ER, Donegan E, Mosley JW. Role of viral load in heterosexual transmission of human immunodeficiency virus type 1 by blood transfusion recipients. Transfusion Safety Study Group. Am J Epidemiol. 1997 Oct 15;146(8):655-61. doi: 10.1093/oxfordjournals.aje.a009331. PMID 9345119
- [Background] Vasil'eva VF, Vorob'eva KP. [Study of magnesium transport in the dog kidney by the method of stopping urine emission in chronic experiments]. Fiziol Zh SSSR Im I M Sechenova. 1975 Jan;61(1):130-5. No abstract available. Russian. PMID 1109967
- [Background] Wilkinson DA, Operskalski EA, Busch MP, Mosley JW, Koup RA. A 32-bp deletion within the CCR5 locus protects against transmission of parenterally acquired human immunodeficiency virus but does not affect progression to AIDS-defining illness. J Infect Dis. 1998 Oct;178(4):1163-6. doi: 10.1086/515675. PMID 9806051
- Available data/document: Study Protocol: TSS — http://biolincc.nhlbi.nih.gov/studies/tss/ — Samples and characterization data. NHLBI provides controlled access to samples through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a materials use agreement.